CLINICAL TRIAL: NCT05516784
Title: Impact of CYP2C19 Genotype-guided Clopidogrel and Ticagrelor Treatment on Platelet Function Test and Metabolomics Profile Among Coronary Artery Disease (CAD) Patients Undergoing Percutaneous Coronary Intervention (PCI)
Brief Title: Impact of CYP2C19 Genotype-guided Clopidogrel and Ticagrelor Treatment on Platelet Function Test and Metabolomics Profile
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Mohammed Rezeq Akkaif, Principle investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 56795
Record Dates: First submitted 2022-08-23; First posted 2022-08-26 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Coronary Artery Disease (CAD)
MeSH Terms: conditions — Coronary Artery Disease | interventions — Clopidogrel; Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Clopidogrel (Active Comparator): The primary endpoint is the non-inferiority in platelet reactivity of clopidogrel versus ticagrelor among CYP2C19*2 or *3 allele carriers.
  Interventions: Drug: Clopidogrel; Drug: Ticagrelor
- Ticagrelor (Experimental): The primary endpoint is the non-inferiority in platelet reactivity of clopidogrel versus ticagrelor among CYP2C19 CYP2C19*2 or *3 allele carriers.
  Interventions: Drug: Clopidogrel; Drug: Ticagrelor

INTERVENTIONS:
Drug: Clopidogrel — Comparison of platelet reactivity between clopidogrel and ticagrelor
  Other Names: Plavix
Drug: Ticagrelor — Comparison of platelet reactivity between clopidogrel and ticagrelor
  Other Names: Brilinta

SUMMARY:
Several studies have shown that pharmacodynamic (PD) response varies between patients treated with clopidogrel and that individuals with reduced response have an increased risk of recurrent ischemic events, particularly in patients undergoing percutaneous coronary intervention. This is due to several factors influencing the response to clopidogrel, including genetic variations of the cytochrome P450 (CYP) 2C19 enzyme. Loss of function (LOF) carriers of the CYP2C19 gene are associated with the decreased generation of the active metabolite clopidogrel and decreased platelet inhibition, which translates to an increased rate of adverse cardiovascular events, particularly in the setting of percutaneous coronary intervention (PCI). Thus, drug regulatory authorities have cautioned about the decreased efficacy of clopidogrel among individuals with CYP2C19 LOF carriers and suggested using alternative therapies to inhibit p2Y12. Ticagrelor is a new generation P2Y12 receptor inhibitor with greater efficacy for PD and reduced rates of ischemic events compared with clopidogrel and are not affected by the CYP2C19 LOF polymorphism. However, in clinical practice, the genotype-guided selection strategy for the oral P2Y12 inhibitor has been limited despite intensive research efforts. This is due to the interaction of cardiovascular risk factors and molecular and biochemical complications that lead to poor response to platelet inhibitor therapy, which impedes physicians' ability to prescribe a more effective and personalized antiplatelet therapy. Therefore, we must move away from traditional approaches and use integrated systems biology study designs and disciplines to bridge the gap between genotype, phenotype, disease manifestation and/or recurrence. Pharmacometabolomics is a rapidly developing field that takes advantage of a systems pharmacology approach to probe the molecular pathways involved in drug response variability to understand metabolic changes and identify novel biomarkers that can be used to predict response more comprehensively. Using profiles of changes in metabolites can help establish drug exposure fingerprints and clarify the determinants of drug response. This study aims to investigate the Impact of pharmacogenetics-guided clopidogrel and ticagrelor treatment on platelet function test and its association with metabolomics in Coronary Artery Disease (CAD) patients undergoing PCI in Malaysia

ELIGIBILITY:
Inclusion Criteria:

* Males or females.
* Age more than 18 and below 80 years.
* Patients with stable CAD planned for elective PCI.
* Thienopyridine naive for at least two weeks before admission.

Exclusion Criteria:

* Pregnant
* Any urgent/emergent coronary angiography procedure that would not allow for genetic testing to be performed before PCI
* Considered at high risk for bleeding
* History of ischemic or hemorrhagic stroke or transient ischemic attack
* . Current treatment with drugs interfering with CYP3A4 metabolism (to avoid interaction with Ticagrelor): ketoconazole, itraconazole, voriconazole, clarithromycin, nefazodone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir, and telithromycin
* History of ACS within 12 months of screening or need for revascularization
* Any acute or chronic unstable condition.
* Liver disease.
* Have increased bleeding risk, e.g., recent gastrointestinal bleed, uncontrolled high blood pressure, low platelet count.
* History of intolerance or allergy to ticagrelor or clopidogrel
* Patient on dialysis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-08-22 (Actual); Study Completion 2022-08-22 (Actual)

PRIMARY OUTCOMES:
Platelet Reactivity | 4 hours post loading dose
  The primary endpoint is a Platelet reactivity index (PRI) measured by the ELISA-Based Vasodilator-Associated Stimulated Phosphoprotein Phosphorylation Assay 4hours/hospital discharge post randomization to clopidogrel vs ticagrelor. Vasodilator-stimulated phosphoprotein (VASP) measurement is the most specific approach to evaluate the extent to which P2Y12 receptors are functionally blocked by a P2Y12 antagonist.

SECONDARY OUTCOMES:
Participants With Any Event From the Composite of All-cause Mortality, and MI | Randomization up to 30 days
  Participants with death from any cause or MI. If no event, censoring occurs at the earliest of patient withdrawal of consent or date of the scheduled withdrawal from therapy
Participants With MI Event | Randomization up to 30 days
  Participants with MI event. If no event, censoring occurs at the earliest of patient withdrawal consent or date of scheduled withdrawal from therapy
Participants With Major or Minor Bleeding | First dosing up to 30 days
  Participants with major (fatal/life-threatening or other) or minor bleed based on need for treatment, number of transfusions, hemoglobin decrease, and other factors

CONTACTS AND LOCATIONS:
Overall Officials: Baharudin Ibrahim, Principal Investigator — Faculty of Pharmacy, University of Malaya, Kuala Lumpur 50603, Federal Territory Malaysia; Nur Aizati Athirah Daud, Principal Investigator — School of Pharmaceutical Sciences, Universiti Sains Malaysia, Penang 11800, Malaysia; Mohammed Ahmed Akkaif, Principal Investigator — School of Pharmaceutical Sciences, Universiti Sains Malaysia, Penang 11800, Malaysia; Muhammed Ali Sk Abdul Kader, Principal Investigator — Department of Cardiology, Penang General Hospital, Penang 10990, Malaysia
Locations (1):
- Department of Cardiology, Penang General Hospital, George Town, Pulau Pinang, Malaysia

REFERENCES:
- [Background] Akkaif MA, Daud NAA, Sha'aban A, Ng ML, Abdul Kader MAS, Noor DAM, Ibrahim B. The Role of Genetic Polymorphism and Other Factors on Clopidogrel Resistance (CR) in an Asian Population with Coronary Heart Disease (CHD). Molecules. 2021 Apr 1;26(7):1987. doi: 10.3390/molecules26071987. PMID 33915807
- [Background] Akkaif MA, Sha'aban A, Daud NAA, Yunusa I, Ng ML, Sk Abdul Kader MA, Noor DAM, Ibrahim B. Coronary Heart Disease (CHD) in Elderly Patients: Which Drug to Choose, Ticagrelor and Clopidogrel? A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Cardiovasc Dev Dis. 2021 Sep 30;8(10):123. doi: 10.3390/jcdd8100123. PMID 34677192
- [Derived] Akkaif MA, Daud NAA, Noor DAM, Sha'aban A, Kader MASA, Ibrahim B. The Impact of CYP2C19 Genotype on the Platelet Reactivity Index (PRI) among Chronic Coronary Syndromes (CCS) Patients Undergoing Percutaneous Coronary Intervention (PCI): Affectability of Rapid Genetic Testing. Cardiovasc Drugs Ther. 2025 Apr;39(2):347-356. doi: 10.1007/s10557-024-07544-6. Epub 2024 Jan 15. PMID 38224415